CLINICAL TRIAL: NCT04484688
Title: Perindopril+Bisoprolol in Therapy of Patients With Atrial Fibrilation
Brief Title: Prestilol(Perindopril+Bisoprolol) in Therapy of Patients With Atrial Fibrilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aversi Clinic (Other)
Responsible Party: Principal Investigator, David Maisuradze, MD,FESC, Aversi Clinic
Other Study IDs: Prestilol
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Patient Participation
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: perindopril-bisoprolol — outpatients with permanent atrial fibrillation and with preserved ejection fraction
  Other Names: prestilol

SUMMARY:
The study aims to evaluate the effectiveness and safety of oral fixed-dose combination of bisoprolol/perindopril in patients with permanent atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:permanent atrial fibrillation with normal EF -

Exclusion Criteria:AF with decreased EF

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with AF and normal EF
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
12-ecg and echocardiography evaluation after 1 month treatment | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Aversi Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR